CLINICAL TRIAL: NCT03970785
Title: Intraoperative Fluorescence of Gangliogliomas and Neuroepithelial Dysembryoplastic Tumors
Brief Title: Intraoperative Fluorescence of Ganglogliomas and Neuroepithelial Dysembryoplastic Tumors
Acronym: FLUOGOD
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_3046_FLUOGOD
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Surgical Procedure, Unspecified
Keywords: fluorescein; gangliogliomas; glioneuronal; Dysembryoplastic Neuroepithelial Tumor
MeSH Terms: conditions — Ganglioglioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
One of the key issues of tumour brain surgeries is to clearly define the borders of the tumor. The investigators proposed to evaluate the feasibility of intraoperative fluorescein guidance. Patients will be identified from the list of patients operated on under fluorescence to collect clinical datas. Surgical videos will be analyzed to assess the presence of intraoperative fluorescence and its subjectively judged intensity. MRI data will be extracted from the radiological reports to assess quality extraction. No additional data will be produced

DETAILED DESCRIPTION:
Gangliogliomas typically present as a slow-growing, cystic mass taking contrast, while dysembryoplastic neuro-epithelial tumors commonly show microcystic patterns, inconstant contrast-enhancement and are preferentially located on the internal face of the temporal lobe. The cornerstone of the treatment of these two entities remains surgery, as it provides good oncological outcomes and control of seizures. Surgical resection keeps a major role for these tumors. Thus, one of the key issues is to clearly define the borders of the tumor during surgery, a point of considerable importance for these curable lesions. Then, the investigators proposed to evaluate the feasibility of intraoperative fluorescein guidance, a technique based on the staining of blood-brain barrier breakdown areas with fluorescein. Patients will be identified from the list of patients operated on under fluorescence maintained by the department since the acquisition of the technique. Clinical datas will be collected and surgical videos will be analyzed to assess the presence of intraoperative fluorescence and its subjectively judged intensity (absent, weak, medium, strong). MRI data (quality of excision: total, subtotal or partial according to usual criteria) will be extracted from the radiological reports. No additional data will be produced

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old patient
* Fluoroguided removal of a histologically proven Ganglioglioma or Dysembryoplastic Neuroepithelial Tumors between 2015-2018
* Surgical video available

Exclusion Criteria:

* Absence of surgical video
* Adults who are subject to legal protection (protection of justice, guardianship, guardianship)
* Patient objecting to the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seven patients (5 men, 2 women, mean age 30 year-old) underwent fluorescein-guided resection of gangliogliomas (5/7; 4 WHO Grade I, 1 WHO Grade III) and DNT (2/7).
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Number of Intraoperative tumor fluorescence | 2 months
  Number of patients which present intraoperative tumor fluorescence. Fluorescence will be assessed using surgical videos.

SECONDARY OUTCOMES:
Number of allergic events | 2 months
  Number of allergic events during fluorescein-based surgery
Percentage of excised tumour volume | 2 months
  Percentage of excised tumour volume. Quality of excision on the post-operative MRI control according to the volume of the remaining pathological contrast intake (complete, subtotal or partial)
Number of epilepsy events after surgery | 2 months
  Occurence of postoperative epilepsy events using Engels classification. (Class I: Free of disabling seizures, Class II: Rare disabling seizures ("almost seizure-free"), Class III: Worthwhile improvement, Class IV: No worthwhile improvement)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Jean LE RESTE, Md, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU Rennes, Rennes, France